CLINICAL TRIAL: NCT03168997
Title: Memantine Treatment in Alzheimer's Disease Patients Stratified With Behavioral and Psychological Symptoms of Dementia (BPSD) Symptoms and Cognitive Severity: A Multi-center, Open-label, Parallel-group and Prospective Clinical Study
Brief Title: Memantine Treatment in Alzheimer's Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Cuibai (Other)
Responsible Party: Sponsor-Investigator, Wei Cuibai, Professor, MD, PhD., Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17237T
Record Dates: First submitted 2017-05-16; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease Memantine
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild AD (Other): Memantine Hydrochloride 20mg tablet per day by mouth on mild AD
  Interventions: Drug: Memantine Hydrochloride
- Moderate AD (Other): Memantine Hydrochloride 20mg tablet per day by mouth on moderate AD
  Interventions: Drug: Memantine Hydrochloride
- Severe AD (Other): Memantine Hydrochloride 20mg tablet per day by mouth on severe AD
  Interventions: Drug: Memantine Hydrochloride

INTERVENTIONS:
Drug: Memantine Hydrochloride — Memantine Hydrochloride treatment according to clinical routine treatment
  Other Names: Memantine

SUMMARY:
The aim of this study is to investigate whether there will be any efficacy difference of Memantine treatment in different cognitive severity AD patients stratified with BPSD

DETAILED DESCRIPTION:
Planed to enroll a total of 222 patients with mild, moderate or severe AD treated with Memantine in 2017-2018 from 15 centers.

ELIGIBILITY:
Inclusion Criteria:

1. Probable AD based on the diagnosis criteria of NIA-AA guideline (the U.S. National Institute on Aging and Alzheimer's Association guideline, McKhann et al, 2011[8];
2. Male or female, 50 years and older ;
3. All inpatients or outpatients recruited into this study must meet MMSE score ≤24 points, patients with MMSE score as 21-24 points will be enrolled into mild group, patients with MMSE score as 10-20 points will be enrolled into moderate group, patients with MMSE score less than 10 points will be enrolled into severe group.
4. Have a reliable caregiver who can accompany the patient to the site to complete the required study procedures;
5. Provide the informed consent.

Exclusion Criteria:

1. Patients with disturbance of consciousness of any causes;
2. Patients with severe aphasia or physical disability who were unable to complete neuropsychological examination;
3. Patients with mental illness;
4. Patients with a history of alcoholism and drug addiction, or traumatic brain injury, epilepsy, encephalitis, normal-pressure hydrocephalus and other neurological disorders causing cognitive impairment;
5. Patients with systemic diseases causing dementia (e.g. liver and kidney insufficiency, endocrine disorders, vitamin deficiency);
6. Patients with a history of ischemic or hemorrhagic cerebrovascular diseases, and vascular diseases (stroke foci) as confirmed by imaging examination;
7. Subjects who are unwilling or unable to abide by the study requirement.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog change | ADAD-cog Change from baseline to 24 weeks
  Alzheimer's Disease Co-operative Study Alzheimer's Disease Assessment Scale - cognitive section is the cognitive evaluation scale

IPD SHARING:
Plan to Share IPD: Undecided